CLINICAL TRIAL: NCT03149653
Title: A Prospective, Randomized, Controlled, Double-blind, Crossover-Design, Mono-center, Phase IV Study Comparing the Effect of Omegaven in Combination With Clinoleic or Lipoplus or SMOFlipid in Home Parenteral Nutrition Patients
Brief Title: Crossover Study on the Effect of Omegaven in Combination With Different Lipid Emulsions in Home Parenteral Nutrition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Collaborators: Charles University, Czech Republic (Other); Ministry of Health, Czech Republic (Other Government)
Responsible Party: Principal Investigator, Frantisek Novak, Chief physician, General University Hospital, Prague
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NT13236-4/2012
Record Dates: First submitted 2017-04-11; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Parenteral Nutrition
Keywords: lipid emulsion; olive oil; fish oil; intestinal failure; home parenteral nutrition
MeSH Terms: conditions — Hyperphagia; Intestinal Failure | interventions — ClinOleic; BaseLine dental cement; fish oil triglycerides; SMOFlipid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 Home Parenteral Nutrition, Cross-over (Experimental): Random Cycle Sequence - Cycle 1: Clinoleic (baseline), 50g/per day, 42 days Clinoleic + Omegaven, 40g + 10g/per day, 28 days. Cycle 2: Lipoplus (baseline), 50g/per day, 42 days Lipoplus + Omegaven, 40g + 10g/per day, 28 days. Cycle 3: SMOFlipid (baseline), 50g/per day, 42 days SMOFlipid + Omegaven, 40g + 10g/per day, 28 days.
  Interventions: Drug: ClinOleic (baseline); Drug: ClinOleic + Omegaven; Drug: Lipoplus (baseline); Drug: Lipoplus + Omegaven; Drug: SMOFlipid (baseline); Drug: SMOFlipid + Omegaven
- 2 Home Parenteral Nutrition, Cross-over (Active Comparator): Random Cycle Sequence - Cycle 1: Clinoleic (baseline), 50g/per day, 42 days Clinoleic + Omegaven, 40g + 10g/per day, 28 days. Cycle 2: Lipoplus (baseline), 50g/per day, 42 days Lipoplus + Omegaven, 40g + 10g/per day, 28 days. Cycle 3: SMOFlipid (baseline), 50g/per day, 42 days SMOFlipid + Omegaven, 40g + 10g/per day, 28 days.
  Interventions: Drug: ClinOleic (baseline); Drug: ClinOleic + Omegaven; Drug: Lipoplus (baseline); Drug: Lipoplus + Omegaven; Drug: SMOFlipid (baseline); Drug: SMOFlipid + Omegaven
- Comparator3 (No Intervention): Healthy Control

INTERVENTIONS:
Drug: ClinOleic (baseline) — Lipid emulsion in pharmacy compounded all-in-one admixture
  Other Names: ClinOleic 20% Baxter
  Arms: 1 Home Parenteral Nutrition, Cross-over; 2 Home Parenteral Nutrition, Cross-over
Drug: ClinOleic + Omegaven — Lipid emulsion in pharmacy compounded all-in-one admixture
  Other Names: ClinOleic 20% Baxter + Omegaven 10% Fresenius Kabi
  Arms: 1 Home Parenteral Nutrition, Cross-over; 2 Home Parenteral Nutrition, Cross-over
Drug: Lipoplus (baseline) — Lipid emulsion in pharmacy compounded all-in-one admixture
  Other Names: Lipoplus 20% BBraun Melsungen
  Arms: 1 Home Parenteral Nutrition, Cross-over; 2 Home Parenteral Nutrition, Cross-over
Drug: Lipoplus + Omegaven — Lipid emulsion in pharmacy compounded all-in-one admixture
  Other Names: Lipoplus 20% BBraun Melsungen + Omegaven 10% Fresenius Kabi
  Arms: 1 Home Parenteral Nutrition, Cross-over; 2 Home Parenteral Nutrition, Cross-over
Drug: SMOFlipid (baseline) — Lipid emulsion in pharmacy compounded all-in-one admixture
  Other Names: SMOFlipid 20% Fresenius Kabi
  Arms: 1 Home Parenteral Nutrition, Cross-over; 2 Home Parenteral Nutrition, Cross-over
Drug: SMOFlipid + Omegaven — Lipid emulsion in pharmacy compounded all-in-one admixture
  Other Names: SMOFlipid 20% Fresenius Kabi + Omegaven 10% Fresenius Kabi
  Arms: 1 Home Parenteral Nutrition, Cross-over; 2 Home Parenteral Nutrition, Cross-over

SUMMARY:
The aim of this study was to evaluate the safety and tolerance of ClinOleic or Lipoplus or SMOFlipid lipid emulsions. After 6 weeks of each lipid emulsion, Omegaven (fish oil) was added for a further 4 weeks. The safety and tolerance was evaluated after each lipid emulsion cycle by biochemistry, hematology and coagulation variables, vital signs and adverse events. We also analysed fatty acid profiles in plasma or erythrocyte phospholipids, antioxidant enzyme activities, lipid peroxidation products, plasma lipids and pro-inflammatory cytokine production after in vitro stimulation of whole blood by lipopolysacharide in HPN patients. The non-interventional group of healthy controls was included for comparison.

DETAILED DESCRIPTION:
Intravenous lipid emulsions (LEs) are an indispensable part of home parenteral nutrition (HPN). All commercially obtainable LEs are applicable for HPN in providing a source of energy and essential fatty acids. The originally used soyabean oil-based LE (Intralipid) have been suspected of being associated with a higher risk of pro-inflammatory lipid-mediator production due to their high content of n-6 polyunsaturated fatty acids. The more modern mixes of soyabean oil, and/or olive oil, and/or fish oil LEs with beneficial responses compared with Intralipid are available. Given that there are no clear clinical recommendations for LE application in HPN, we performed this cross-over design, phase 4 study comparing ClinOleic, Lipoplus or SMOFlipid in chronic intestinal failure patients with additional escalation of fish oil using Omegaven.

ELIGIBILITY:
Inclusion Criteria:

* Home parenteral nutrition patients in need of parenteral nutrition administration > 4 days/week
* Parenteral duration expectancy > 8 months
* Stable clinical condition without any complications in the past 2 months
* Written consent from the subject

Exclusion Criteria:

* Known hypersensitivity to any of the active substances or excipients
* Unstable conditions
* Active cancer or its treatment
* Established immunodeficiency
* Advanced organ dysfunction from chronic disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01-15 (Actual); Primary Completion 2016-01-07 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline lipid emulsion production of TNF-alpha after in vitro stimulation of whole blood by lipopolysacharide at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The whole blood culture supernatant concentration of TNF-alpha (ng/L)
Change from baseline lipid emulsion production of IL-1-beta after in vitro stimulation of whole blood by lipopolysacharide at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The whole blood culture supernatant concentration of IL-1-beta (ng/L)
Change from baseline lipid emulsion production of IL-6 after in vitro stimulation of whole blood by lipopolysacharide at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The whole blood culture supernatant concentration of IL-6 (ng/L)
Change from baseline lipid emulsion production of IL-8 after in vitro stimulation of whole blood by lipopolysacharide at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The whole blood culture supernatant concentration of IL-8 (ng/L)

SECONDARY OUTCOMES:
Change from baseline lipid emulsion plasma concentration of TNF-alpha at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration of TNF-alpha (ng/L)
Change from baseline lipid emulsion plasma concentration of IL-1-beta at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration of IL-1-beta (ng/L)
Change from baseline lipid emulsion plasma concentration of IL-6 at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration of IL-6 (ng/L)
Change from baseline lipid emulsion plasma concentration of IL-8 at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration of IL-8 (ng/L)
Change from baseline lipid emulsion plasma concentration ratio of oxidized LDL/LDL cholesterol at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration ratio of oxidized LDL/LDL cholesterol (ox-LDL/LDL-C)
Change from baseline lipid emulsion plasma concentration of triglycerides at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration of triglycerides (mmol/L)
Change from baseline lipid emulsion plasma concentration of total cholesterol at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration of total cholesterol (mmol/L)
Change from baseline lipid emulsion plasma concentration of HDL cholesterol at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration of HDL cholesterol (mmol/L)
Change from baseline lipid emulsion plasma concentration of LDL cholesterol at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration of LDL cholesterol (mmol/L)
Change from baseline lipid emulsion plasma phospholipid fatty acid profile at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma phospholipid fatty acid profile (mol%)
Change from baseline lipid emulsion erythrocyte phospholipid fatty acid profile at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The erythrocyte phospholipid fatty acid profile (mol%)
Change from baseline lipid emulsion plasma concentration of fibrothelial growth factor 19 at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma concentration of fibrothelial growth factor 19 (ng/L)
Change from baseline lipid emulsion erythrocyte superoxide dismutase activity at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The erythrocyte activity of SOD (U/g Hb)
Change from baseline lipid emulsion erythrocyte catalase activity at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The erythrocyte activity of CAT (U/g Hb)
Change from baseline lipid emulsion erythrocyte glutathione peroxidase activity at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The erythrocyte activity of GPX (U/g Hb)
Change from baseline lipid emulsion erythrocyte glutathione reductase activity at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The erythrocyte activity of GR (U/g Hb)
Change from baseline lipid emulsion plasma paraoxonase 1 activity at 4 weeks of Omegaven lipid emulsion addition | day 42, day 70
  The plasma activity of PON1 (U/L)
Alteration of liver function | week 6, week 10, week 16, week 20, week 26, week 30
  Liver function tests
Septic complications | week 6, week 10, week 16, week 20, week 26, week 30
  Catheter-related bloodstream infections

CONTACTS AND LOCATIONS:
Overall Officials: Frantisek Novak, MD, PhD, Principal Investigator — General University Hospital, Prague
Locations (1):
- General University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No